CLINICAL TRIAL: NCT05318352
Title: The Effect of Using Transcranial Direct Current Stimulation in Improving Quality of Sleep in Athletes: A Randomized Controlled Trial
Brief Title: tDCS in Improving Quality of Sleep in Athletes
Acronym: tDCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Alia A. Alghwiri, Professor of Physiotherapy, University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 80-2021
Record Dates: First submitted 2022-03-04; First posted 2022-04-08 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Sleep Disorder
Keywords: tDCS, Sleep, Athletes
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial Direct Current Stimulation (tDCS) (Experimental): Athletes with poor sleep quality will receive tDCS over the right and left prefrontal cortex (F3 and F4 areas) with a constant current of 1.5 mA intensity that lasts for 20 minutes, 3 times a week for 2 weeks in daytime.
  Interventions: Device: Transcranial Direct Current Stimulation
- Sham transcranial Direct Current Stimulation (tDCS) (Sham Comparator): Athletes with poor sleep quality will receive sham tDCS over the right and left prefrontal cortex.
  Interventions: Device: Transcranial Direct Current Stimulation

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation — Transcranial direct current stimulation (tDCS) is a noninvasive brain stimulation technique that modulates cortical activity. tDCS has been conducted to improve wide range of neurological impairments including sleep.

SUMMARY:
Sleep disturbances in athletes was found prevalent and affect their cognitive and physical abilities and increase the risk of injury. Moreover, studies showed also that a better sleep produces a better athletic performance. Therefore, it is important to find out management strategies that improve quality of sleep in this population.

Transcranial direct current stimulation (tDCS) is a noninvasive brain stimulation technique that modulates cortical activity. tDCS has been conducted to improve wide range of neurological impairments including sleep. tDCS was used in improving the quality of sleep in older adults and in athletes. Both studies found improvement in some sleep indices.

DETAILED DESCRIPTION:
Research ethics:

1. Institutional Review Board approval was sought out from University of Jordan before the beginning of the study.
2. Informed consent will be obtained from athletes guaranteed their approval to participate in the study.
3. To insure the privacy of participants, every athlete will be assigned a study identification number.
4. All results will be stored in a locked cabinet/computer.

Study design and participants:

This is double -blinded randomized placebo-controlled parallel trial. The study will be reported according to the Consolidated Standards of Reporting Trials (CONSORT) statement for non-pharmacological treatment (Boutron et al., 2008). Data will be collected prospectively from athletes from different sports in Jordan.

Sample Size calculation:

The sample size was calculated using G*Power software, according to the study of Acler et al,. 2013. The study found Cohen d=0.7012 effect size of transcranial direct current stimulation on PSQI. Based on 0.7012 effect size, bidirectional alpha of 0.05, and 80% test power, a minimum of 70 participants were needed to the study. The sample will be increased by 20 % to compensate possible dropouts, overall sample of 84 participants will be included in this study.

Procedures:

1. Eligible athletes will be approached via the Jordanian Olympic Committee to participate in this study.
2. A researcher will explain the whole procedures of the research study including the randomization.
3. Athletes will go through baseline assessment.
4. A randomization will be conducted using a computerized program.
5. Participants will be invited to start the intervention sessions.
6. At the end of the treatment, athletes will go through post-treatment assessment.

The demographic data will be collected from eligible participants by a blinded assessor at baseline period. The included participants will be randomly allocated to tDCS groups or control group by a website (www.randomization.com) in a balanced allocation ratio. Outcome measures will be conducted by an assessor blinded to group randomization at baseline, after tDCS interventions, and at 1-month follow up. Allocation will be concealed from the assessor until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Athletes who are 12 years of age and older.
* Athletes who have a complaint of sleep impairment determined by >5 total score on Pittsburg Sleep Quality Index (PSQI).

Exclusion Criteria:

* Athletes who is using sleep medications or treatment.
* Athletes who have more than 1 concussion in the past year.
* Wearing a pacemaker.
* Pregnant athletes.
* Athletes who have repetitive migraine
* Athletes who are wearing a metal implant.
* Athletes who have epilepsy.

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Severity of sleep impairment (using Insomnia Severity Index) | Baseline.
  The total score ranges between 0 and 28 with a higher score indicates more sever insomnia (worse).
Severity of sleep impairment (using Insomnia Severity Index) | After 4 weeks.
  The effect of the intervention on insomnia severity. The total score ranges between 0 and 28 with a higher score indicates more sever insomnia (worse).
Quality of Sleep (using Actigraph activity monitor) | Baseline.
  The wGT3X-BT is ActiGraph's flagship activity monitor, used to capture and record continuous, high resolution physical activity and sleep/wake information.
Quality of Sleep (using Actigraph activity monitor) | After 3 weeks.
  The effect of the intervention on quality of sleep. The wGT3X-BT is ActiGraph's flagship activity monitor, used to capture and record continuous, high resolution physical activity and sleep/wake information.
Daytime sleepiness (using Epworth Sleepiness Scale) | Baseline.
  It consists of 8 items where the subject uses a 4-point Likert scale to rate how likely they would be to fall asleep in 8 different scenarios of daily activities. The total score ranges between 0-24 with a higher score indicates worse daytime sleepiness.
Daytime sleepiness (using Epworth Sleepiness Scale) | After 4 weeks.
  The effect of the intervention on daytime sleepiness. It consists of 8 items where the subject uses a 4-point Likert scale to rate how likely they would be to fall asleep in 8 different scenarios of daily activities. The total score ranges between 0-24 with a higher score indicates worse daytime sleepiness.
The Quality of sleep (Using Pittsburgh Sleep Quality Index) | Screening for eligibility.
  The total score ranges from 0 to 21 with a higher score indicates poor quality of sleep (worse). A cut-off score of >5 indicates poor sleep quality.
The Quality of sleep (Using Pittsburgh Sleep Quality Index) | After 4 weeks.
  The effect of the intervention on the Quality of sleep. The total score ranges from 0 to 21 with a higher score indicates poor quality of sleep (worse). A cut-off score of >5 indicates poor sleep quality.
The Quality of sleep (Using Pittsburgh Sleep Quality Index) | After 2 Months from baseline.
  The effect of the intervention on the Quality of sleep. The total score ranges from 0 to 21 with a higher score indicates poor quality of sleep (worse). A cut-off score of >5 indicates poor sleep quality.

SECONDARY OUTCOMES:
The Quality of Life (using Medical Outcomes Study Short Form 12) | Baseline.
  The effect of the intervention on Quality of Life. The total score ranges between 0% to 100% with higher score indicates a better quality of life (better).
The Quality of Life (using Medical Outcomes Study Short Form 12) | After 4 weeks.
  The effect of the intervention on Quality of Life. The total score ranges between 0% to 100% with higher score indicates a better quality of life (better).
The severity of anxiety, depression, and stress (using Depression Anxiety Stress Scale-21) | Baseline.
  The effect of the intervention on anxiety, depression, and stress. The total score ranges from 0 to 63 with higher score indicates more severe anxiety, depression, and stress (worse).
The severity of anxiety, depression, and stress (using Depression Anxiety Stress Scale-21) | After 4 weeks.
  The effect of the intervention on anxiety, depression, and stress. The total score ranges from 0 to 63 with higher score indicates more severe anxiety, depression, and stress (worse).

CONTACTS AND LOCATIONS:
Overall Officials: Alia Alghwiri, PhD, Principal Investigator — University of Jordan
Locations (1):
- University of Jordan, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Etoom M, Alwardat M, Alghwiri A, Lena F, Romigi A. Effects of Transcranial Direct Current Stimulation on Sleep in Athletes: A Protocol of a Randomized Controlled Trial. J Clin Med. 2022 Oct 5;11(19):5883. doi: 10.3390/jcm11195883. PMID 36233749